CLINICAL TRIAL: NCT00152828
Title: A Phase I/II Trial of the Cyclooxygenase-2 Inhibitor Celecoxib in the Treatment of Patients With Locally Advanced Carcinoma of the Cervix
Brief Title: Celebrex - Cervix: Celecoxib in the Treatment of Patients With Locally Advanced Carcinoma of the Cervix
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: NCIC Clinical Trials Group (Network); Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 00-0431-C; National Cancer Instit.Canada
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Cervix Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Celecoxib (Experimental): Celecoxib
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib

SUMMARY:
This is a phase I/II study to evaluate the safety and toxicity of celecoxib in combination with standard concurrent cisplatin and radiotherapy in women with locally advanced cervix cancer. In addition, we aim to determine the effect of celecoxib (Celebrex) on tumour oxygenation, interstitial fluid pressure, COX-2 levels, prostaglandin E2 levels, angiogenesis and apoptosis.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven carcinoma of the cervix, with visible/palpable tumours; FIGO stage T1B-3B, NO/1, MO, to be treated with definitive radiotherapy and chemotherapy
* ECOG performance status of 0, 1, or 2
* Adequate hematologic function; Granulocyte count greater than 1.5 x 109/L, Platelet count greater than 100 x 109/L
* Adequate organ function; Serum creatinine £ 1.25 x ULN, or a calculated creatinine clearance ³ 50 mL/min, Serum bilirubin £ 1.25 x ULN and AST/ALT £ 3xULN
* No prior treatment for cervix cancer
* Informed consent

Exclusion Criteria:

* Use of an NSAID in the 2 weeks prior to study enrollment
* Patients with an active malignancy at another site
* Patients with significant cardiac, renal, or pulmonary disease or any other medical conditions that may preclude radical therapy
* Patients who have significant history of ischaemic heart disease or stroke who would be deemed not suitable for cessation of their daily prophylactic aspirin
* Patients with history of peptic ulcer disease or previous NSAID related gastrointestinal bleeding
* Patients with hypersensitivity to NSAIDS or celecoxib, or sulfonamides
* Patients who unwilling or unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2001-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety - Tolerance of concurrent celecoxib with standard cisplatin/radiotherapy | 1 year

SECONDARY OUTCOMES:
Objective changes in tumour oxygenation and IFP | 1 year
Objective molecular marker response (COX-2, PGE2, VEGF, apoptosis) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Fyles, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada